CLINICAL TRIAL: NCT00885989
Title: A Placebo-Controlled, Combined Single and Multiple Rising Dose Study to Determine the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SLV338 After Intravenous Administration in Healthy Male Subjects
Brief Title: Safety and Tolerability of the First IV Dosing of SLV338 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Responsible Party: Ellis Ides, Solvay Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S338.1.002; 2008-006753-40
Record Dates: First submitted 2009-01-30; First posted 2009-04-22 (Estimated); Last update posted 2010-01-29 (Estimated); Status verified 2010-01

CONDITIONS: Healthy
Keywords: SLV338; phase I; healthy volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: SLV338
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SLV338 — 5 - 1000 mg IV
  Arms: 1
Drug: Placebo — Placebo
  Arms: 2

SUMMARY:
This study will investigate the safety and tolerability of the first IV dosing of SLV338 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* healthy

Exclusion Criteria:

* not healthy

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2009-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability parameters, including administration site tolerability, adverse events, clinical laboratory tests, vital signs and ECG | 7 days

SECONDARY OUTCOMES:
Pharmacokinetic parameters: AUC, Cmax, tmax, t½, λz, CL, CLR, Vz, Vss, MRT, Ae, and fe. | 48 hours
Pharmacodynamic parameters: Plasma levels of ANP, cGMP, BNP, VIP, Big ET, ET-1, angiotensin II and aldosteron. Urinary volume and urine levels of cGMP, sodium, potassium, chloride, uric acid and creatinine, and creatinine clearance. | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (1):
- Site 1, London, United Kingdom